CLINICAL TRIAL: NCT01431430
Title: Prospective Double Blind Multicentre Randomized Trial of Vitamine D Estimating the Profit of a Treatment by Vitamin D3 at the Dose of 100000 UI by Comparison With a Treatment in the Dose of 12 000 UI at Renal Transplanted Patients
Brief Title: VITamine D Supplementation in RenAL Transplant Recipients - VITALE
Acronym: VITALE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire Crinex (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P100103
Record Dates: First submitted 2011-08-22; First posted 2011-09-09 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Renal Transplant Candidate for Right Kidney
Keywords: Vitamine D; renal transplantation; diabetes mellitus; cancer; cardiovascular complications
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol 100 000 UI (Experimental): Cholecalciferol 100 000 UI FORTHIGHTLY for 2 months then monthly for 22 months
  Interventions: Drug: Cholecalciferol 100 000 UI
- Cholecalciferol 12 000 UI (Control) (Active Comparator): Cholecalciferol 12 000 UI FORTHIGHTLY for 2 months then monthly for 22 months.
  Interventions: Drug: Cholecalciferol 12 000 UI

INTERVENTIONS:
Drug: Cholecalciferol 100 000 UI — Cholecalciferol 100 000 UI FORTHIGHTLY for 2 months then monthly for 22 months
  Arms: Cholecalciferol 100 000 UI
Drug: Cholecalciferol 12 000 UI — Cholecalciferol 12 000 UI FORTHIGHTLY for 2 months then monthly for 22 months.
  Arms: Cholecalciferol 12 000 UI (Control)

SUMMARY:
It has been proposed that the intake of high dose of cholecalciferol may have beneficial non classical effects (beside bone health). This could include the reduction of type 2 diabetes mellitus, cardiovascular diseases, cancers, autoimmune and infectious diseases. These pleiotropic effects are mostly documented by observational and experimental studies or small intervention trials. In renal transplant recipients, vitamin D insufficiency, defined as circulating 25(OH)vitamin D (25OHD) less than 30 ng/mL, is a frequent finding and this population is at risk of the previously cited complications.The primary purpose of this study is to compare the effects of high dose vs. low dose of cholecalciferol on a composite endpoint consisting in de novo diabetes mellitus, cardiovascular diseases, de novo cancer and patient death.Renal transplant recipients between 12 and 48 months after transplantation will be randomized to blindly receive either high or low dose of cholecalciferol with a follow-up of 2 years.

DETAILED DESCRIPTION:
Rationale :

Vitamin D cannot be considered any more as only necessary to prevent rickets or osteomalacia. Calcitriol produced in the kidney is known to have classical endocrine PHOSPHOCALCIC properties. More recently, vitamin D has been shown to play an important role in reducing the risk of many chronic diseases including type 2 diabetes mellitus, cardiovascular diseases, cancers, autoimmune and infectious diseases. These effects may be secondary to local production of calcitriol and to its autocrine and paracrine actions on cellular proliferation and differentiation, apoptosis, insulin and renin secretion, interleukin and bactericidal proteins production. These pleiotropic effects are mostly documented by observational and experimental studies or small intervention trials that most often evaluated intermediate parameters. In renal transplant recipients, vitamin D insufficiency (circulating 25OHD<30 ng/mL or 75 nmol/L) , is a frequent finding with more than 80% of patients displaying this profile.

Objective:

Primary objective: compare the effects of high dose vs. low dose of cholecalciferol on a composite endpoint including

* De novo diabetes mellitus (fasting glycemia > 7 MMOLES/l or glycemia > 11 MMOLES/l)
* Cardiovascular complications (acute coronary heart disease, acute heart failure, lower-extremity arterial disease, cerebrovascular disease).
* De novo cancer,
* Patient death.

Secondary objectives : compare the effects of high dose vs. low dose of cholecalciferol on

* The occurrence of each event constituting the primary endpoint
* Blood pressure and blood pressure control (number and dosage of antihypertensive drugs)
* Echocardiography findings
* Infection including opportunistic (CMV, pneumocystis, nocardial infection, cryptococcal infection, aspergillosis)
* Acute rejection episode
* Renal allograft function including estimated glomerular filtration rate and proteinuria - Graft survival
* PHOSPHOCALCIC biological and clinical relevant parameters : Evolution of serum 25OHD, calcaemia, phosphataemia, serum PTH, bone mineral density and incidence of fractures
* Renal lithiasis

Study protocol

Number of patients: 320 patients in each group Inclusions : 2 years Follow-up after inclusion : 2 years Prospective, randomized, multicentre, double blind clinical study comparing high dose cholecalciferol [100 000 UI FORTHIGHTLY for 2 months then monthly for 22 months) vs. low dose cholecalciferol [12 000 UI FORTHIGHTLY for 2 months then monthly for 22 months).

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients between 12 and 48 months after transplantation with a stable renal function during the past 3 months.
* Vitamine D insufficiency defined as a concentration of 25OHD lower than 30 ng/ml.
* Patient between 18 and 75 years old
* Patient capable of understanding the advantages and the risks of the study.
* Affiliated with social security health insurance
* Written informed consent

Exclusion Criteria:

* Calcaemia > 2,7 mmol/l
* Phosphataemia > 1,5 mmol/l
* Serum creatinine > 250 µmol/l
* Treatment by an active form of the vitamin D not being able to be interrupted
* Transplant of an organ other than the kidney
* Type I or type II diabetes mellitus
* Past medical history of granulomatosis or active granulomatosis
* Primary hyperoxaluria
* Malabsorption proved by the liposoluble vitamins
* Simultaneous participation in another therapeutic essay
* Patients presenting a drug addiction or a psychiatric disorder
* Pregnant or breast-feeding women
* Vitamin D hyper sensibility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-02-02 (Actual)

PRIMARY OUTCOMES:
De novo diabetes mellitus | 2 years
  De novo diabetes mellitus (fasting glycemia > 7 mmoles/l or glycemia > 11 mmoles/l)
Cardiovascular complications | 2 years
  Cardiovascular complications (acute coronary heart disease, acute heart failure, lower-extremity arterial disease, cerebrovascular disease).
De novo cancer | 2 years
  Diagnosis of the incidence of any new cancer
Patient death | 2 years

SECONDARY OUTCOMES:
Blood pressure control | 2 years
  Blood pressure and blood pressure control (number and dosage of antihypertensive drugs)
Echocardiography findings | 2 years
  Comparison of left ventricular ejection fraction
Infection including opportunistic | 2 years
  Infection including opportunistic (CMV, pneumocystis, nocardial infection, cryptococcal infection, aspergillosis)
Acute rejection episode | 2 years
Renal allograft function | 2 years
  Renal allograft function including estimated glomerular filtration rate, proteinuria
Graft survival | 2 years
Phosphocalcic biological and clinical relevant parameters | 2 years
  PHOSPHOCALCIC biological and clinical relevant parameters : Evolution of serum 25OHD, calcaemia, phosphataemia, serum PTH, bone mineral density and incidence of fractures
Renal lithiasis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric THERVET, MD, PhD, Principal Investigator — European Georges Pompidou Hospital
Locations (1):
- Georges Pompidou European Hospital, Paris, France

REFERENCES:
- [Background] Courbebaisse M, Bourmaud A, Souberbielle JC, Sberro-Soussan R, Moal V, Le Meur Y, Kamar N, Albano L, Thierry A, Dantal J, Danthu C, Moreau K, Morelon E, Heng AE, Bertrand D, Arzouk N, Perrin P, Morin MP, Rieu P, Presne C, Grimbert P, Ducloux D, Buchler M, Le Quintrec M, Ouali N, Pernin V, Bouvier N, Durrbach A, Alamartine E, Randoux C, Besson V, Hazzan M, Pages J, Colas S, Piketty ML, Friedlander G, Prie D, Alberti C, Thervet E. Nonskeletal and skeletal effects of high doses versus low doses of vitamin D3 in renal transplant recipients: Results of the VITALE (VITamin D supplementation in renAL transplant recipients) study, a randomized clinical trial. Am J Transplant. 2023 Mar;23(3):366-376. doi: 10.1016/j.ajt.2022.12.007. Epub 2023 Jan 9. PMID 36695682
- [Background] Courbebaisse M, Alberti C, Colas S, Prie D, Souberbielle JC, Treluyer JM, Thervet E. VITamin D supplementation in renAL transplant recipients (VITALE): a prospective, multicentre, double-blind, randomized trial of vitamin D estimating the benefit and safety of vitamin D3 treatment at a dose of 100,000 UI compared with a dose of 12,000 UI in renal transplant recipients: study protocol for a double-blind, randomized, controlled trial. Trials. 2014 Nov 6;15:430. doi: 10.1186/1745-6215-15-430. PMID 25376735